CLINICAL TRIAL: NCT05765825
Title: Phase II, Single-Arm Study of Low-Dose Radiotherapy (LDRT) Concurrent Cisplatin/Carboplatin Plus Etoposide With Serplulimab for Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Study of Low-Dose Radiotherapy Concurrent Chemotherapy With Serplulimab for Patients With ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPUR
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; Carboplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT concurrent cisplatin/carboplatin + etoposide + serplulimab (Experimental): Participants will receive the following treatment regimens: The induction period consists of 4 cycles of 21 days each. Low-dose radiotherapy(LDRT) at 15Gy/5f will be performed concurrently from Day 1 to Day 5 (D1-D5) of Cycle 1. An efficacy assessment will be performed at the end of Cycle 2. For patients with primary lung lesions (intrathoracic lesions) evaluated as small PR (tumor shrinkage < 80%)/SD/PD, ldrt at 15Gy/5f will be performed in addition to serplulimab with chemotherapy in Cycle 3. For subjects evaluated as PD/SD/PR with extrathoracic residual metastases, ldrt at 15Gy/5f will be performed in addition to serplulimab with chemotherapy in Cycle 4. After the induction period, the subjects will continue to receive maintenance treatment with serplulimab.
  Interventions: Drug: serplulimab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide; Radiation: Thoracic radiation therapy (TRT)

INTERVENTIONS:
Drug: serplulimab — Serplulimab will be administered by intravenous infusion at a dose of 4.5mg/kg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, and clinical status.
  Other Names: HLX10
Drug: Cisplatin — Cisplatin will be administered as intravenous infusion at a dose of 75 mg per meter squared (75 mg/m^2) after completion of serplulimab on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: Cisplatin injection
Drug: Carboplatin — Carboplatin will be administered as intravenous infusion at a dose of area under the concentration-time curve (AUC) of 5 mg/mL/min on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: Carboplatin injection
Drug: Etoposide — Etoposide will be administered intravenously at a dose of 100 mg/m^2 on Days 1, 2 and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: Etoposide injection
Radiation: Thoracic radiation therapy (TRT) — Participants will receive concurrent low-dose radiotherapy treatment, in once daily fractions, 3 Gy per fraction, to a target dose of 15 Gy in 5 fractions from Day 1-Day 5 in the first cycle, third cycle（ For patients with primary lung lesions (intrathoracic lesions) evaluated as small PR (tumor shrinkage < 80%)/SD/PD），forth cycle（for subjects evaluated as PD/SD/PR with extrathoracic residual metastases).
  Other Names: low-dose radiotherapy

SUMMARY:
This is a Phase II, single arm, multicenter study designed to evaluate the safety and efficacy of low-dose radiotherapy (LDRT) concurrent cisplatin/carboplatin plus etoposide with serplulimab in participants who have extensive-stage small cell lung cancer (ES-SCLC) and are chemotherapy-navïe for their extensive-stage disease.

DETAILED DESCRIPTION:
Enrolled patients will receive the following treatment regimen: LDRT-concurrent cisplatin/carboplatin plus etoposide in combination with serplulimab. The induction period consists of 4 cycles of 21 days each. Low-dose radiotherapy at 15Gy/5f will be performed concurrently from Day 1 to Day 5 (D1-D5) of Cycle 1. An efficacy assessment will be performed at the end of Cycle 2 and one week before the start of Cycle 3. For patients with primary lung lesions (intrathoracic lesions) evaluated as small PR (tumor shrinkage < 80%)/SD/PD, low-dose radiotherapy at 15Gy/5f will be performed in addition to serplulimab with chemotherapy in Cycle 3. For subjects evaluated as PD/SD/PR with extrathoracic residual metastases, low-dose radiotherapy at 15Gy/5f will be performed in addition to serplulimab with chemotherapy in Cycle 4. Definition of extrathoracic lesions for radiotherapy: Metastases to liver, metastases to adrenals and metastases to lymph nodes (at the discretion of the investigator).

After the induction period, the subjects will continue to receive maintenance treatment with serplulimab. Prophylactic cranial irradiation (PCI) is allowed for treatment according to local standard of care. Patients will be treated until loss of clinical benefit, unacceptable toxicity, withdrawal of informed consent, or death, whichever occurs first.

ELIGIBILITY:
Main Inclusion Criteria:

1. Histologically or cytologically confirmed ES-SCLC
2. No prior treatment for ES-SCLC
3. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation.
4. ECOG performance status of 0 or 1
5. Life expectancy >= 3 months
6. Adequate hematologic and end-organ function
7. For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
8. Negative human immunodeficiency virus (HIV) test at screening
9. Negative hepatitis B surface antigen (HBsAg) test at screening
10. Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following: Negative total hepatitis B core antibody (HBcAb), or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test. The HBV DNA test will be performed only for participants who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
11. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for participants who have a positive HCV antibody test.
12. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception
13. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Main Exclusion Criteria:

1. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
2. Participants with pulmonary artery invasion
3. History of leptomeningeal disease
4. Uncontrolled tumor-related pain
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
6. Uncontrolled or symptomatic hypercalcemia
7. Active or history of autoimmune disease or immune deficiency
8. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
9. Active tuberculosis
10. Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
11. History of malignancy other than small cell lung cancer (SCLC) within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to approximately 24 months
  The time from the date of first dosing of serplulimab to the first appearance of objective disease progression (according to RECIST1.1) or death from any cause (if it occurs before disease progression).

SECONDARY OUTCOMES:
PFS Rate at 6 Months and 1 Year | Baseline up to 1 year
  PFS rate at 6 months and 1 year, defined as the proportion of patients who have not experienced disease progression or death from any cause at 6 months and 1 year separately, as determined by the investigator according to RECIST v1.1.
Overall Survival (OS) | Baseline up to approximately 24 months
  The time from the date of first dosing of serplulimab to death from any cause.
OS Rate at 1 Year and 2 Years | Baseline to 2 years or death, whichever occurs first.
  OS rate at 1 year and 2 years, defined as the proportion of patients who have not experienced death from any cause at 1 year and 2 years.
Duration of response (DOR) | Baseline to disease progression or death from any cause (whichever occurs first)(up to approximately 24 months)
  defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Disease control rate (DCR) | Baseline up to approximately 24 months
  defined as the proportion of participants who have a best overall response of CR or PR or stable disease (SD), as determined by the investigator according to RECIST v1.1.
Percentage of Participants With Adverse Event | Baseline up to approximately 36 months
  • The incidence and severity of adverse events, with severity determined according to the U.S. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAEv5.0)

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Study Chair — West China Hospital
Locations (8):
- China (8):
  - Chongqing University cancer hospital, Chongqing, Chongqing Municipality
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - LiaoNing Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - China West Hospital, Chengdu, Sichuan
  - GuiZhou Provincial People's Hospital, Guiyang

IPD SHARING:
Plan to Share IPD: No